CLINICAL TRIAL: NCT01624909
Title: The China PEACE (Patient-centered Evaluative Assessment of Cardiac Events) Prospective Study of Acute Myocardial Infarction
Brief Title: China PEACE-Prospective AMI Study
Status: Completed | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Collaborators: Ministry of Health, China (Other Government)
Responsible Party: Sponsor
Other Study IDs: WSGY-201202025-3
Record Dates: First submitted 2012-06-17; First posted 2012-06-21 (Estimated); Last update posted 2015-08-31 (Estimated); Status verified 2015-08

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A venous blood sample of 20mL will be collected at 1-month visit and 12-month visit for biomarker analysis and storage for future genetic studies;
  A urine samples of 40mL will be collected at 1-month visit and 12-month visit for biomarker analysis and storage.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Coronary heart disease (CHD) and heart attacks pose a serious health risk to men and women, however little information is available about how evidence-based therapies are incorporated appropriately into routine clinical practice in China. In addition, basic data and evidence about safety and efficacy of treatment for AMI is limited. By consecutively recruiting AMI patients in 40 hospitals of different levels, this study will examine various real-life factors, that may affect patients recovery after a heart attack. Practical guidelines and risk model for AMI patients will be established based on the findings, to improve patients outcomes in future finally.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is a major concern in public health globally, as well as in China, and AMI is one of the leading causes of mortality and morbidity. Remarkable variations of resources available and health system performance have been noted, however little information is available about how evidence-based therapies are incorporated appropriately into routine clinical practice in China. In addition, basic data and evidence about safety, efficacy, and effectiveness of treatment for AMI during long-term recovery is limited. Practical and applied knowledge from large unselected population is needed to guide practice and policy for quality improvement and cost reduction.

This study will enroll patients with a confirmed diagnosis of AMI consecutively in 20 tertiary hospitals and 20 secondary hospitals scattered all over China. At study entry, participants will be interviewed during their index hospitalization, to collect information about symptoms, functioning, quality of life, and medical care. Demographic characteristics, medical history, clinical features, diagnostic tests, medications, procedures, and in-hospital outcomes of patients will be abstracted from medical records by well trained professional abstractors. At 1 month, 6 month, and 12 month after discharge, participants will return to the clinic for follow up visits, a face-to-face interview will be conducted to get information about clinical events, symptoms, functioning, quality of life, and medical care during the recovery period. At 1-Month and 12-Month follow-up visit, blood and urine sample will be collected. Participants' blood samples will be stored for future biologic and genetic studies. This study will examine various real-life factors that may affect patients recovery after a heart attack, including patients' characteristics and treatment measures. Practical guidelines, quality evaluative system, and risk model for AMI patients will be established based on the findings, to improve patients outcomes in future finally.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients with acute myocardial infarction according to positive cardiac biomarkers (Troponin I/T, CK-MB or CK≥ local laboratory upper limit of normal values within 24 hours after initial presentation, and at least one of the following two supporting evidence of ischemia (ischemic symptoms occurring within 24 hours before admission or up to 72 hours for STEMI; ECG changes indicative of new ischemia).

Exclusion Criteria:

* Previously enrolled in the PEACE study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In 40 hospitals of different levels in China, 4000 hospitalized patients with acute myocardial infarction will be enrolled consecutively.
Sampling Method: Non-Probability Sample
Enrollment: 4286 (Actual)
Dates: Start 2012-12; Primary Completion 2014-05 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiovascular events (MACE) | 1 year
  Composite of major adverse cardiovascular events (MACE) including cardiac death, non-fatal AMI, coronary revascularization procedure, or ischemic stroke.

SECONDARY OUTCOMES:
Symptoms status (SAQ) | 1 year
Quality of life (EQ-5D) | 1 year
Depression (PHQ-8) | 1 year
Stress (PSS-4) | 1 year
Cardiac death | 1 year
Fatal or non-fatal AMI | 1 year
Coronary revascularization procedure | 1 year
Ischemic stroke | 1 year
Re-admission | 1 year
Adherence to medications for secondary prevention | 1 year
  Taking the following medications for 6 or more days per week: aspirin, clopidogrel, ACEI/ARB, statin and beta-blockers
Control of risk factors | 1 year
  Control of hypertension, diabetes, dyslipidemia, smoking, and obesity

OTHER OUTCOMES:
Cognitive function (MMSE) | 1 year
Sexual activity/function | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Lixin Jiang, M.D., Ph.D., Principal Investigator — China National Center for Cardiovascular Diseases; Harlan M Krumholz, M.D., S.M., Principal Investigator — Yale University
Locations (1):
- Fuwai Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Li J, Dharmarajan K, Bai X, Masoudi FA, Spertus JA, Li X, Zheng X, Zhang H, Yan X, Dreyer RP, Krumholz HM. Thirty-Day Hospital Readmission After Acute Myocardial Infarction in China. Circ Cardiovasc Qual Outcomes. 2019 May;12(5):e005628. doi: 10.1161/CIRCOUTCOMES.119.005628. PMID 31092023
- [Derived] Shang P, Liu GG, Zheng X, Ho PM, Hu S, Li J, Jiang Z, Li X, Bai X, Gao Y, Xing C, Wang Y, Normand SL, Krumholz HM. Association Between Medication Adherence and 1-Year Major Cardiovascular Adverse Events After Acute Myocardial Infarction in China. J Am Heart Assoc. 2019 May 7;8(9):e011793. doi: 10.1161/JAHA.118.011793. PMID 31057004
- [Derived] Huo X, Khera R, Zhang L, Herrin J, Bai X, Wang Q, Lu Y, Nasir K, Hu S, Li J, Li X, Zheng X, Masoudi FA, Spertus JA, Krumholz HM, Jiang L. Education level and outcomes after acute myocardial infarction in China. Heart. 2019 Jun;105(12):946-952. doi: 10.1136/heartjnl-2018-313752. Epub 2019 Jan 19. PMID 30661037
- [Derived] Jiang Z, Dreyer RP, Spertus JA, Masoudi FA, Li J, Zheng X, Li X, Wu C, Bai X, Hu S, Wang Y, Krumholz HM, Chen H; China Patient-centered Evaluative Assessment of Cardiac Events (PEACE) Collaborative Group. Factors Associated With Return to Work After Acute Myocardial Infarction in China. JAMA Netw Open. 2018 Nov 2;1(7):e184831. doi: 10.1001/jamanetworkopen.2018.4831. PMID 30646375
- [Derived] Guan W, Venkatesh AK, Bai X, Xuan S, Li J, Li X, Zhang H, Zheng X, Masoudi FA, Spertus JA, Krumholz HM, Jiang L. Time to hospital arrival among patients with acute myocardial infarction in China: a report from China PEACE prospective study. Eur Heart J Qual Care Clin Outcomes. 2019 Jan 1;5(1):63-71. doi: 10.1093/ehjqcco/qcy022. PMID 29878087
- [Derived] Qi Y, Wang W, Zhang K, An S, Wang S, Zheng J, Tang YD. Development and validation of Women Acute Myocardial Infarction in-Hospital Mortality Score (WAMI Score). Int J Cardiol. 2018 May 15;259:31-39. doi: 10.1016/j.ijcard.2017.12.010. PMID 29579607